CLINICAL TRIAL: NCT02706990
Title: In Vivo Kinematic Analysis of Total Knee Replacement With a Kinematic Retaining or a Posterior Stabilized Design During Activities of Daily Living
Brief Title: Fluoroscopic Analysis of Total Knee Replacement With a Kinematic Retaining or a Posterior Stabilized Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: K-10
Record Dates: First submitted 2016-03-07; First posted 2016-03-11 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2016-09

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physica KR (Other): Patients who have received a Physica KR total knee implant.
  Interventions: Device: Physica KR
- Physica PS (Other): Patients who have received a Physica PS total knee implant.
  Interventions: Device: Physica PS

INTERVENTIONS:
Device: Physica KR — Kinematic retaining total knee implant
  Arms: Physica KR
Device: Physica PS — Posterior stabilized total knee implant
  Arms: Physica PS

SUMMARY:
The aim of this study is to evaluate the in vivo kinematics of TKA performed with two different prosthesis: a kinematic retaining (Physica KR) and a posterior-stabilized (Physica PS) design by means of fluoroscopic analysis during activities of daily living (rising from a chair, stairs climbing, leg extension). In comparison with asymptomatic knee. Patterns of femoral rollback will be analyzed to assess if they are motor-task dependent and correlated with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients submitted to Total knee arthroplasty (TKA) with Physica KR or PS;
2. Patients with an appropriate initial fixation and stability of the knee prosthesis;
3. Patients achieving a minimum flexion of 100° or a Knee Society Score (KSS) ≥ 65 (fair/good postoperative outcome) at 6-month follow-up;
4. Patients affected by primary or secondary Osteoarthritis (OA) before surgery;
5. Patients who understand the requirements of the study and are willing and able to comply with activities required for fluoroscopic examination;
6. Patients who have signed the Ethics Committee approved study-specific Informed Consent Form.

Exclusion Criteria:

1. Patients with misalignment or axial malrotation of the knee prosthesis;
2. Patients not able to achieve a minimum flexion of 100° or with a KSS Knee Score ≤ 65 points at 6-month follow-up;
3. Patients who had or have planned a surgery on their uninvolved knee within a year;
4. Muscular insufficiency or absence of muscololigamentous supporting structures required for adequate soft tissue balance;
5. Patients who have significant neurological or musculoskeletal disorders or disease that may adversely affect gait and compromise functional recovery and evaluation;
6. Patients who have neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device;
7. Any psychiatric illness that would prevent comprehension of the details and nature of the study;
8. Participation in any experimental drug/device study within the 6 months prior to the screening visit
9. Female patients who are pregnant, nursing, or planning a pregnancy due to x-rays exposition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the roll-back mechanism measured with the tibio-femoral contact points at different degrees of flexion | 6 months
  Using a software to replicate the movement using Computer-aided design (CAD) models. The movement is studied and the distance made by the femur on the tibia is calculated giving the information of the roll back.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marega, MD, Principal Investigator — Ospedale San Camillo, Trento
Locations (1):
- Ospedale San Camillo, Trento, Trento, Italy